CLINICAL TRIAL: NCT06444230
Title: Effects Of Routine Physical Therapy With And Without Neuro-Developmental Technique On Gross Motor Function, Spasticity And Health Related Quality Of Life In Diplegic Cerebral Palsy- A Randomized Controlled Trail
Brief Title: Effects of Routine Physical Therapy With and Without Neurodevelopmental Technique on GMF, Spasticity and HRQOL in Diplegic CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Shehzeena Ashraf, Principal Investigator, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-UOL-536-09-2023
Record Dates: First submitted 2024-05-29; First posted 2024-06-05 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; gross motor function; neurodevelopmental technique; health realted quality of life; routine physical therapy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuro-developmental Physical Therapy+ Routine Physical Therapy (Experimental): * Protocol of 40 minutes focusing on gross motor functional movements including upright sitting at the table, walking, kneeling, running and stair climbing.
  * Used a Neuro-developmental method to inhibit undesirable movement patterns and facilitate favorable movement patterns.
  * Weight-bearing exercises that involved proprioceptive training while in various positions (such as quadruped, kneeling, half kneeling, and standing).
  * Facilitating weight transfer forward, backward, and sideways during balancing reactions from various balance board postures
  Interventions: Other: Routine Physical therapy with Neurodevelopmental technique; Other: Routine Physical therapy
- Routine Physical therapy: (Experimental): All children in this group received physical therapy of 40 minutes, 3 times per week for 12weeks, which included passive stretching with focus on diplegic limb 8 minutes, neck and trunk postural control for 8 minutes, strength training 8 minutes, ambulation and gait training for 8 minutes with 2 minutes rest interval between each set of exercise.
  Interventions: Other: Routine Physical therapy with Neurodevelopmental technique; Other: Routine Physical therapy

INTERVENTIONS:
Other: Routine Physical therapy with Neurodevelopmental technique — participants will recieve a session of 40 minutes including routine physical therapy along with the neurodevelopmental technique for 3 times a week for 12 weeks
Other: Routine Physical therapy — participants will recieve a session of 40 minutes including, stretching, neck and trunk stabilization and strengthening exercise followed by a warm up and cool down for 3 times a week for 12 weeks follo

SUMMARY:
The aim of this study is to investigate the effects of routine physical therapy with and without neurodevelopmental technique on gross motor function, spasticity and health related quality of life in diplegic cerebral palsy.

DETAILED DESCRIPTION:
The neurological illness known as cerebral palsy is caused by damage to the growing brain and therefore is indicated by anomalies of muscle strength, mobility, and motor functions. Cerebral palsy affects posture, muscle tone, and movement development. Neurodevelopmental technique and routine physical therapy are considered to be effective in treatment of cerebral palsy. This study will investigate the combined effects of neurodevelopmental technique and routine physical therapy versus routine physical therapy on gross motor function, spasticity, and health related quality of life in diplegic cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an age of 8 to 18 years of both genderswith confirm diagnosis of diplegic cerebral palsy
* Patients could ambulate functionally
* Patients having limited or no prior exposure to NDT
* Individuals with mild to moderate diplegic cerebral palsy, based on established classification scales (GMFM grade I-III)

Exclusion Criteria:

* Patients with other motor or sensory dysfunctions and unable to understand and obey commands
* Patient undergone any orthopedic surgery that was ought to treatspasticity
* Patients with spasticity level 4-5 according to Modified Ashworth Scale
* Patients with Botulinum toxins type A injection within last 6 months

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale | 9 months
  UMN syndrome's component of spasticity is an increase in muscular stretch out reflexes that is velocity-dependent and accompanied by an increase in muscle tone. Bryan Ashworth developed the Ashworth Scale in 1964 while treating patients with MS as a way to grade spasticity. The original Ashworth scale, which rated spasticity on a scale of 0 to 4, classified it as either having no resistance or having limbs that were stiff in flexion or extension. They added 1+ to the scale to boost sensitivity(Bohannon & Smith, 1987). Muscle spasticity is rated using the modified Ashworth scale score ranging from 0 to 4, having total 6 grades
Gross Motor Function Measure | 9 months
  Each item is rated on a four-point ordinal system of assessment. A score of 0 means the task cannot be performed, a score of 1 means the task is able to be started (10% completion), a score of 2 means the task may be completed partially (10% to 100% completion), and a score of 3 means the task is capable of being finished.Every unobserved item on the GMFM-88 receives a score of 0. On the contrast, GMFM-66, however, items that were not seen received a "not tested" or "missing" score.Both versions of GMFM has an excellent reliability
Cerebral Palsy Quality of Life Questionnaire for Children and Adolescent | 9 months
  The Cerebral Palsy Quality of Life for Children (CP QOL-Child) is the very first quality of life survey founded on the International Classification of Function (ICF) created particularly for kids with CP.The CP QOL-Child is available in two versions: the main caregiver-proxy report version (proxy version) for kids ages 4 to 12 and a self-report version for kids ages 9 to 12. The CP QOL-Child's internal consistency, test-retest reliability, and construct validity have all been proven to be reliable and valid.

SECONDARY OUTCOMES:
Manual Muscle Testing | 9 months
  The most popular technique for identifying muscle strength deficits is MMT. According to the dimensions of the muscle and the power of the examiner, scores range from zero contractions to a contraction which can be done against gravity and can withstand the examiner's "maximal" resistance. The examiner rates the muscular groups under study as either "weak" or "strong" on a scale of zero to five while applying force against the participant's resistance

CONTACTS AND LOCATIONS:
Overall Officials: Shehzeena Ashraf, Study Chair — University of Lahore
Locations (1):
- University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No